CLINICAL TRIAL: NCT01664559
Title: Pain Control for Intrauterine Device Placement: A Randomized, Double Blind Control Trial of Ketorolac Prior to Intrauterine Device Placement.
Brief Title: Pain Control for Intrauterine Device Placement: A Trial of Ketorolac Prior to Intrauterine Device Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lynn Ngo (Other)
Responsible Party: Sponsor-Investigator, Lynn Ngo, Resident Physician, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WRHR 5K12001259-12 - toradol
Record Dates: First submitted 2012-06-28; First posted 2012-08-14 (Estimated); Results first posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-11

CONDITIONS: Pain Control With IUD Insertion
Keywords: intrauterine device; ketorolac; toradol; mirena; paragard; pain control
MeSH Terms: conditions — Agnosia | interventions — Ketorolac; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo with 1cc normal saline IM (Placebo Comparator): If the patient is randomized to the placebo arm, they will receive 1cc of normal saline via the intramuscular route.
  Interventions: Drug: Normal Saline
- Toradol, 30mg in 1cc IM (Experimental): If the patient is randomized to the toradol (ketorolac) arm, they will receive 30mg of toradol in a 1cc volume via the intramuscular route.
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — Ketorolac 30mg intramuscular injection, 1cc volume
  Other Names: Brand name: toradol; Serial # (01) 1 030409 379649 7
  Arms: Toradol, 30mg in 1cc IM
Drug: Normal Saline — Placebo arm, 1cc of normal saline, 0.9%, intramuscular injection
  Other Names: REF# 196604
  Arms: Placebo with 1cc normal saline IM

SUMMARY:
Intrauterine device (IUD) placement can be painful for patients during and after the procedure. Fear of pain from IUD insertion can be a barrier to obtaining this highly effective long acting reversible contraception. Currently there are no proven effective methods for reduction of pain during and after placement of modern IUDs (Mirena IUD and Paragard IUD). Ketorolac has not been studied in regards to decreasing pain during and after IUD insertion although it is used by some providers for this purpose. It is a strong NSAID that is indicated for the treatment of moderate acute pain. In the intramuscular form it has an analgesia onset of action at 30min, thus may be a plausible option for pain management in the office setting compared to oral NSAIDs, which have a longer time to onset of analgesia and have not been proven to be effective in reducing pain associated with IUD placement. The primary aim of this study is to determine whether ketorolac (Toradol) decreases pain associated with intrauterine device placement compared to placebo. We hypothesize that administration of ketorolac 30mg intramuscularly at least 30 minutes prior to IUD insertion will decrease pain scores by at least 20mm on a visual analog scale at various time points during IUD insertion when compared to placebo of normal saline injection.

DETAILED DESCRIPTION:
Modern intrauterine devices are highly effective long acting reversible forms of contraception. The Mirena IUD is 99.8% effective and the Paragard copper IUD is 99.2% effective in preventing pregnancy (Zieman 2010). Fear of intrauterine device placement can be a barrier to obtaining this highly effective form of birth control. The current standard of care for pain management during and after IUD placement is no medication, as randomized control trials published to date have limited data regarding use of medications to decrease pain. There has been one trial to suggest that the use of naproxen with 1% lidocaine paracervical block compared to paracervical block alone may decrease pain after IUD placement in primarily nulliparous patients. However, this study was with the much wider and no longer available Dalkon Shield IUD. In addition, this study did not show any significant decrease in pain scores during IUD placement (Massey 1974). Studies to evaluate effectiveness of motrin and misoprostol have shown no significant decrease in pain scores during and after IUD insertion, although the majority of participants in these studies were multiparous (Jensen 1998, Hubacher 2006, Saav 1997). There is some suggestion that 2% lidocaine gel one minute prior to IUD insertion may have some decrease in pain, although this study was poorly designed (Oloto 1996).

There have been no studies published to date regarding the use of ketorolac for decreasing pain during and after IUD placement. Ketorolac is an acetic acid NSAID that reversibly inhibits COX 1 and 2, leading to decreased formation of prostaglandin precursors, and is indicated for the use of moderate acute pain in the short term setting. Its administration in the office setting may be good option for providers since intramuscular administration leads to analgesia beginning at 30 minutes, maximal effect 1 to 2 hours after administration, and duration of analgesia approximately 4 to 6 hours for the 30mg intramuscular injection.

Although there is no standard of care in regards to pain medication administration prior to IUD placement, providers at UCSD often suggest certain options. These include ibuprofen at least one hour prior to the procedure, or ibuprofen taken within a few hours after the procedure, or ketorolac injection at least 15-30 minutes prior to the procedure. It would be beneficial for providers to have an evidence based option for patients.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous and multiparous women ages 18-50, who are English or Spanish speaking, who present for intrauterine device placement for contraception or menorrhagia (in the case of Mirena IUD insertion).

Exclusion Criteria:

* Pregnancy
* Any diagnosed chronic pain issues (i.e. fibromyalgia, endometriosis, dysmenorrhea, irritable bowel syndrome, interstitial cystitis)
* If the patient has taken any pain medications within 6 hours of enrollment, including aspirin or other NSAIDs
* Misoprostol administration within 24 hours of enrollment
* History of prior IUD insertion
* Known allergy to NSAIDs including diagnosis of aspirin or NSAID induced asthma or urticaria
* Known contraindications to NSAIDs, such as the following medications that are risk category D (consider therapy modification) or X (avoid combination) including

  * bile acid sequestrants (D - may decrease absorption of NSAIDs)
  * cyclosporine (D - NSAIDs may enhance the nephrotoxic effects)
  * drotrecogin alfa (D - NSAIDs may enhance the adverse/toxic effects, cause bleeding)
  * floctafenine (X - may enhance adverse/toxic effect of NSAIDs)
  * lithium (D - NSAIDs may decrease serum concentration)
  * methotrexate (D - NSAIDs may decrease excretion)
  * pentoxifylline (X - Ketorolac may enhance adverse/toxic effects)
  * probenecid (X - may increase serum concentration of Ketorolac)
  * rivaroxaban (D - Anti-platelet drugs may enhance anti-coagulation effect)
  * SSRIs (D - may enhance the anti-platelet effect of NSAIDs, NSAIDs may diminish the therapeutic effect of SSRIs)
  * warfarin (D - NSAIDs may enhance the anti-coagulation effect)
* Renal insufficiency (by history and/or chart review)
* Peptic ulcer disease or history of significant gastrointestinal bleeding
* Known thrombocytopenia, known coagulopathy, or known bleeding disorder
* Known contraindications to IUD

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2012-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn L Ngo, MD, Study Director — University of California, San Diego; Sheila Mody, MD MPH, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

REFERENCES:
- [Background] Allen RH, Bartz D, Grimes DA, Hubacher D, O'Brien P. Interventions for pain with intrauterine device insertion. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD007373. doi: 10.1002/14651858.CD007373.pub2. PMID 19588429
- [Background] Roche NE, Li D, James D, Fechner A, Tilak V. The effect of perioperative ketorolac on pain control in pregnancy termination. Contraception. 2012 Mar;85(3):299-303. doi: 10.1016/j.contraception.2011.10.001. Epub 2011 Nov 30. PMID 22133656
- [Background] Edelman AB, Schaefer E, Olson A, Van Houten L, Bednarek P, Leclair C, Jensen JT. Effects of prophylactic misoprostol administration prior to intrauterine device insertion in nulliparous women. Contraception. 2011 Sep;84(3):234-9. doi: 10.1016/j.contraception.2011.01.016. Epub 2011 Mar 3. PMID 21843686
- [Derived] Ngo LL, Ward KK, Mody SK. Ketorolac for Pain Control With Intrauterine Device Placement: A Randomized Controlled Trial. Obstet Gynecol. 2015 Jul;126(1):29-36. doi: 10.1097/AOG.0000000000000912. PMID 26241253

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo With 1cc Normal Saline IM | Toradol, 30mg in 1cc IM
Started | 34 | 33
Completed | 34 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo With 1cc Normal Saline IM | Toradol, 30mg in 1cc IM | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (5.4) | 26.6 (5.1) | 26.9 (5.3)
Sex/Gender, Customized [Number; unit: female participants] | 34 | 33 | 67
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 13 | 12 | 25
  Hispanic | 4 | 2 | 6
  African American | 14 | 12 | 26
  Asian or Pacific Islander | 1 | 4 | 5
  Other | 2 | 3 | 5
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 27.6 (5.7) | 27.3 (5.8) | 27.4 (5.7)
Gravidity [Median (Inter-Quartile Range); unit: pregnancies] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2]
Parity [Median (Inter-Quartile Range); unit: pregnancies] | 1 [1 to 1] | 1 [1 to 2] | 1 [1 to 1]
Currently breastfeeding [Number; unit: participants] — Not all patients were breastfeeding so this number is not expected to add up to the overall number of baseline participants.
  participants | 15 | 15 | 30
History of loop electrosurgical excision procedure [Number; unit: participants] | 0 | 3 | 3
Level of education [Number; unit: participants] — One participant in the placebo arm did not answer the question about their education status, therefore the sum of the answers for this arm is different than the overall number of baseline participants.
  participants
    Less than high school | 0 | 1 | 1
    High school graduate | 7 | 4 | 11
    Some college | 12 | 11 | 23
    College degree | 7 | 6 | 13
    Graduate degree | 7 | 11 | 18

OUTCOME MEASURES:

1. Primary Outcome: VAS (Visual Analogue Scale) Measurement of Pain
Description: The patient marked their pain on a 0 to 10cm visual analogue scale, where 0 cm is no pain and 10 cm is the worst pain ever.
Time Frame: Pain with IUD placement, measured immediately after placement
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo With 1cc Normal Saline IM | Toradol, 30mg in 1cc IM
Number analyzed (Participants) | 34 | 33
units on a scale | 5.2 [1.2 to 7.4] | 3.6 [1.5 to 6.3]
Statistical Analysis 1: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; Test type: Superiority or Other; p = 0.99, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Pain Scores at Other Time Points During and After IUD Placement
Description: The patient marked their pain on a 0 to 10cm visual analogue scale, where 0 cm is no pain and 10 cm is the worst pain ever.
  1. Prior to injection of study drug, anticipated pain
  2. Pain from study drug injection, measured immediately after injection
  3. Pain from speculum insertion, measured immediately after insertion
  4. Pain with tenaculum placement, measured immediately after placement
  5. Pain with uterine sounding, measured immediately after removal of the sound
  6. Pain at 5 minutes after placement of the intrauterine device
  7. Pain at 15 minutes after placement of the intrauterine device
Time Frame: immediately after each step (see description)
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | Placebo With 1cc Normal Saline IM | Toradol, 30mg in 1cc IM
Number analyzed (Participants) | 34 | 33
cm
  Anticipated pain | 4.4 [1.4 to 6.5] | 3.5 [1.0 to 6.8]
  Pain with injection | 1.0 [0.4 to 2.8] | 0.6 [0.2 to 1.3]
  Speculum insertion | 2.6 [0.6 to 3.7] | 1.5 [0.4 to 3.8]
  Tenaculum placement | 3.9 [2.6 to 5.7] | 2.5 [1.1 to 6.4]
  Uterine sounding | 5.0 [2.5 to 7.5] | 4.3 [1.7 to 7.2]
  5 min after procedure | 2.2 [0.8 to 3.9] | 0.3 [0 to 1.3]
  15 min after procedure | 1.6 [0.4 to 3.6] | 0.1 [0 to 0.9]
Statistical Analysis 1: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; 1) Anticipated pain; Test type: Superiority or Other; p = 0.31, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; 2) pain with injection; Test type: Superiority or Other; p = 0.33, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; 3) speculum insertion; Test type: Superiority or Other; p = 0.72, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; 4) tenaculum placement; Test type: Superiority or Other; p = 0.36, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; 5) uterine sounding; Test type: Superiority or Other; p = 0.64, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; 6) 5 min after placement; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; 7) 15 min after placement; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Nulliparous Patients - Subgroup Analysis
Description: as for outcome 2
Time Frame: immediately after each step (see description)
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | Placebo With 1cc Normal Saline IM | Toradol, 30mg in 1cc IM
Number analyzed (Participants) | 8 | 8
cm
  1) Anticipated pain | 2.8 [0.8 to 5.4] | 3.6 [2.0 to 5.5]
  2) Pain with injection | 1.8 [0.7 to 3.4] | 1.2 [0.8 to 2.7]
  3) Speculum insertion | 2.3 [1.0 to 4.5] | 1.5 [0.3 to 3.1]
  4) Tenaculum placement | 6.3 [3.7 to 7.3] | 4.3 [2.2 to 7.1]
  5) Uterine sounding | 8.4 [6.6 to 9.2] | 6.0 [3.9 to 6.7]
  6) Pain with IUD placement | 8.1 [7.4 to 9.0] | 5.4 [5.0 to 7.4]
  7) 5 min after placement | 3.7 [2.3 to 4.8] | 2.7 [1.5 to 3.3]
  8) 15 min after placement | 4.8 [3.0 to 6.9] | 1.8 [0.2 to 3.2]
Statistical Analysis 1: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; 1) anticipated pain; Test type: Superiority or Other; p = 0.6, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; 2) pain with injection; Test type: Superiority or Other; p = 1.0, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; 3) speculum insertion; Test type: Superiority or Other; p = 0.34, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; 4) tenaculum placement; Test type: Superiority or Other; p = 0.32, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; 5) uterine sounding; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; 6) IUD placement; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; 7) 5 min after placement; Test type: Superiority or Other; p = 0.32, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; 8) 15 min after placement; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Post-insertion Patient Questionnaire
Description: Questions assessed in multiple choice format:
  1. Side effects
  2. injection site pain
  3. overall satisfaction with IUD insertion experience
  4. would they still recommend IUD placement to a friend?
  5. significant pain for which they desired acetaminophen prior to leaving the office?
Time Frame: assessed at 15 minutes after IUD insertion
Measure: Number; unit: participants
Arm/Group | Placebo With 1cc Normal Saline IM | Toradol, 30mg in 1cc IM
Number analyzed (Participants) | 34 | 33
participants
  Reported side effects | 12 | 8
  Injection site pain - just as bad/worse than IUD | 8 | 6
  Satisfied or very satisfied with overall IUD proc | 30 | 31
  Recommend IUD to a friend | 28 | 30
  Desires additional pain medication | 16 | 6
Statistical Analysis 1: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; Reported side effects (nausea, vomiting, dyspepsia, headache, dizziness, drowsiness, injection site itchiness, swelling or pain); Test type: Superiority or Other; p > 0.05, Chi-squared
Statistical Analysis 2: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; Injection site pain (just as bad or worse than IUD procedure); Test type: Superiority or Other; p = 0.76, Chi-squared
Statistical Analysis 3: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; Satisfied or very satisfied with IUD placement procedure; Test type: Superiority or Other; p = 0.76, Chi-squared
Statistical Analysis 4: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; Would recommend IUD placement to a friend; Test type: Superiority or Other; p = 0.35, Chi-squared
Statistical Analysis 5: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; Desires additional pain medication; Test type: Superiority or Other; p = 0.02, Chi-squared

5. Secondary Outcome: Post-insertion Provider Questionnaire
Description: The provider will be asked to fill out a multiple choice format questionnaire:
  1. what level training are you?
  2. which IUD was inserted?
  3. what was the purpose of IUD placement?
  4. what was the position of the uterus?
  5. did the IUD placement process require cervical dilation?
  6. were you able to complete the IUD insertion?
  7. was there bleeding from the cervix that required more than 5 min to control?
  8. were there any major complications with the IUD insertion?
  9. did the patient take tylenol prior to leaving the office?
Time Frame: Immediately after IUD placement, on average within 1 hour
Measure: Number; unit: participants
Arm/Group | Placebo With 1cc Normal Saline IM | Toradol, 30mg in 1cc IM
Number analyzed (Participants) | 34 | 33
participants
  Level of training - PGY1 | 2 | 5
  Level of training - PGY2 | 2 | 13
  Level of training - PGY3 | 3 | 6
  Level of training - PGY4 | 5 | 6
  Level of training - Attending | 1 | 3
  IUD type - levonogestrel | 22 | 28
  IUD type - copper | 12 | 2
  Purpose of IUD - contraception | 33 | 32
  Purpose of IUD - AUB | 1 | 1
  Position of uterus - anteverted | 19 | 20
  Position of uterus - retroverted | 6 | 5
  Position of uterus - midpositioned | 9 | 8
  Cervical dilation needed | 2 | 2
  Able to complete the IUD placement | 34 | 33
  Significant bleeding | 0 | 2
  Major complications | 0 | 0
  Took acetaminophen prior to leaving the office | 17 | 7
Statistical Analysis 1: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; Level of training, PGY 1, 2, 3, 4 and Attending; Test type: Superiority or Other; p = 0.2, Chi-squared
Statistical Analysis 2: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; IUD type (levonorgestrel or copper); Test type: Superiority or Other; p = 0.09, Chi-squared
Statistical Analysis 3: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; Purpose of IUD (contraception or heavy menstrual bleeding); Test type: Superiority or Other; p = 1.0, Chi-squared
Statistical Analysis 4: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; Position of uterus (anteverted, retroverted, midpositioned); Test type: Superiority or Other; p = 0.92, Chi-squared
Statistical Analysis 5: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; Need for cervical dilation; Test type: Superiority or Other; p = 1.0, Chi-squared
Statistical Analysis 6: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; Able to complete the IUD insertion; Test type: Superiority or Other; p = 1.0, Chi-squared, Corrected
Statistical Analysis 7: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; Significant bleeding; Test type: Superiority or Other; p = 0.24, Chi-squared
Statistical Analysis 8: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; Major complications; Test type: Superiority or Other; p = 1.0, Chi-squared
Statistical Analysis 9: Comparison: Placebo With 1cc Normal Saline IM vs Toradol, 30mg in 1cc IM; Took acetaminophen prior to leaving the office; Test type: Superiority or Other; p = 0.02, Chi-squared

ADVERSE EVENTS:
Arm/Group | Placebo With 1cc Normal Saline IM | Toradol, 30mg in 1cc IM
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 0/34 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes